CLINICAL TRIAL: NCT04462094
Title: Comparison of CRP Levels, Neutrophil Count, and Clinical Outcomes of Low Dose Ketamine Between at Anesthesia Induction and at the End of Surgery in Patients Undergo Elective Laparotomy
Acronym: PRO-Ketamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UNUD-CTR-FK260620-002; 1143/UN14.2.2.VII.14/LT/2020 (Other: Committee of Ethical Research of Udayana University)
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: General Anesthesia; Laparotomy; Inflammation
Keywords: stress response; infammation; general anesthesia
MeSH Terms: conditions — Inflammation; Fractures, Stress | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized control trial. It provides a controlled care comparison between low-dose ketamine given at anesthesia induction and at the end-of-surgery.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only care providers involved directly with the subjects in the operating room are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End-of-surgery (Active Comparator): Low-dose ketamine (0.3 mg/kg) in 3 ml normal saline solution given at the end of surgery
  Interventions: Drug: Ketamine 0.3 mg/kg at end-of-surgery; Drug: Ketamine 0.3 mg/kg at anesthesia induction
- Induction (Placebo Comparator): Low-dose ketamine (0.3 mg/kg) in 3 ml normal saline solution given at induction
  Interventions: Drug: Ketamine 0.3 mg/kg at end-of-surgery; Drug: Ketamine 0.3 mg/kg at anesthesia induction

INTERVENTIONS:
Drug: Ketamine 0.3 mg/kg at end-of-surgery — Ketamine 0.3 mg/kg at end-of-surgery (intravenously)
  Other Names: Group E
Drug: Ketamine 0.3 mg/kg at anesthesia induction — Ketamine 0.3 mg/kg at anesthesia induction (intravenously)
  Other Names: Group I

SUMMARY:
The effects of anesthesia and surgery can lead to stress responses that result in hormonal and metabolic changes in the body. The immune system and the nervous system communicate both ways, and it was found that nociception and proinflammatory cytokines play a joint regulatory role, i.e., increased production of proinflammatory cytokines can worsen the pain. Major surgery can trigger the release of cytokines such as IL-1, IL-6, and TNF-α.

DETAILED DESCRIPTION:
The effects of anesthesia and surgery can lead to stress responses that result in hormonal and metabolic changes in the body. The immune system and the nervous system communicate both ways, and it was found that nociception and proinflammatory cytokines play a joint regulatory role, i.e., increased production of proinflammatory cytokines can worsen the pain. Major surgery can trigger the release of cytokines such as IL-1, IL-6, and TNF-α.

The acute analgesic effect of ketamine is generally believed to be mediated through the blockade of the phencyclidine binding site of the N-methyl-d-aspartate (NMDA) receptor of nociceptive neurons. Ketamine can reduce the inflammatory response marked by a decrease in CRP levels to surgical trauma and can prevent secondary damage to tissues/organs that were not initially affected by surgery by reducing inflammation. This also reduces postoperative pain and analgesics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective laparotomy with general anesthesia at Sanglah Hospital from July to September 2020.
2. Patients aged 18-65 years.
3. Patient physical status American American Society of Anesthesiologist (ASA) 1 and 2.

Exclusion Criteria:

1. Contraindication to ketamine.
2. Allergy to morphine
3. Presence of cardiorespiratory chronic diseases.
4. Presence of autoimmune diseases.
5. History of the central nervous system or psychiatric disorders.
6. BMI <18.5 kg/m2 or ≥30 kg/m2.
7. A history of chronic pain killer medications (such as opioid or non-steroidal anti- inflammatory drugs)

Drop Out Criteria

1. Patients with class 3 bleeding during the surgery
2. Patients with more than 5-hours duration of surgery
3. Patients need mechanical ventilation after the surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Serum CRP level | 1-hour before surgery
  Serum C-reactive protein level
Serum CRP level | 24-hours after surgery
  Serum C-reactive protein level
serum neutrophil-count | 1-hour before surgery
  serum neutrophil-count (from a complete blood count test)
serum neutrophil-count | 24-hours after surgery
  serum neutrophil-count (from a complete blood count test)
VAS (visual analog score) | first 24 hours after the surgery
  minimum=0; maximum=10; higher score corresponds to more severe pain
morphine consumption (mg) | first 24 hours after the surgery
  total morphine consumption in 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tjokorda GA Senapathi, Dr, Study Chair — Udayana University; Christopher Ryalino, Dr, Principal Investigator — Udayana University; Made SP Adi, Dr, Study Director — Udayana University
Locations (1):
- Sanglah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No